CLINICAL TRIAL: NCT00070057
Title: An Exploratory, Open-Label Phase I Pharmacodynamic Study of COX-2 Inhibition With Celecoxib (Celebrex) and Aromatase Activity in Breast Cancer
Brief Title: Celecoxib in Treating Postmenopausal Women Who Are Undergoing Surgery for Invasive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01441; NCI-2012-01441 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000329919; MSKCC-03027 (Other: Memorial Sloan-Kettering Cancer Center); N01-CN-35112 (Other: DCP); P30CA008748 (NIH); N01CN35112 (Other Grant/Funding Number: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib

ARMS (3):
- Arm I (celecoxib) (Experimental): Patients receive oral celecoxib twice daily for 1-3 weeks (according to the duration between biopsy and surgery) in the absence of unacceptable toxicity.
  Interventions: Drug: celecoxib; Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (high-dose celecoxib) (Experimental): Patients receive a higher dose of oral celecoxib as in arm I.
  Interventions: Drug: celecoxib; Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm III (surgery) (Active Comparator): Patients do not receive treatment. All patients undergo surgery.
  Interventions: Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: celecoxib — Given orally
  Other Names: Celebrex; SC-58635
  Arms: Arm I (celecoxib); Arm II (high-dose celecoxib)
Procedure: therapeutic conventional surgery — Undergo surgery
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I trial is studying the side effects of celecoxib in treating postmenopausal women with invasive breast cancer who are scheduled to undergo surgery at Memorial Sloan-Kettering Cancer Center. Celecoxib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether celecoxib suppresses aromatase activity in postmenopausal women with invasive breast cancer planning to undergo surgery.

SECONDARY OBJECTIVES:

I. Correlate celecoxib-mediated inhibition of aromatase activity with levels of cyclooxygenase (COX)-2 and HER-2/neu and estrogen receptor status in these patients.

II. Determine the effect of this drug on histology, Ki67, RNA expression profile by microarray analysis, PI3-K, AKT and ERK1/2 MAP kinase activities, and PGE_2 levels in these patients.

III. Determine whether any observed biological effect of this drug is dose-dependent in these patients.

IV. Identify collateral targets (COX-2-independent) of this drug in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 3 treatment arms.

Arm I: Patients receive oral celecoxib twice daily for 1-3 weeks (according to the duration between biopsy and surgery) in the absence of unacceptable toxicity.

Arm II: Patients receive a higher dose of oral celecoxib as in arm I.

Arm III: Patients do not receive treatment.

All patients undergo definitive surgery.

PROJECTED ACCRUAL: A total of 75 patients (25 per treatment arm) will be accrued for this study within 2-3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast carcinoma

  * Tumor at least 1 cm by radiologic estimate or physical exam
  * No disease limited to ductal carcinoma in situ only
* Planning to undergo surgery at Memorial Sloan-Kettering Cancer Center
* Hormone receptor status:

  * Not specified
* Female
* Postmenopausal as defined by at least 1 of the following:

  * No menstrual period within the past 12 months
  * Prior bilateral oophorectomy
* No known liver disease
* No renal insufficiency
* No congestive heart failure
* No coronary artery disease
* No history of documented peptic ulcer disease
* No gastritis
* No medical condition that would preclude definitive surgery
* No allergy to NSAIDs or sulfa-containing drugs
* No connective tissue diseases, including any of the following:

  * Systemic lupus erythematosus
  * Reynaud's disease
  * Scleroderma
* More than 3 months since prior chemotherapy
* More than 2 weeks since prior hormone replacement therapy
* More than 2 weeks since prior tamoxifen
* More than 2 weeks since prior aromatase inhibitors
* More than 2 weeks since prior raloxifene
* More than 2 weeks since prior steroids
* More than 1 week since prior nonsteroidal anti-inflammatory drugs (NSAIDs)
* More than 1 week since prior cyclooxygenase (COX)-2 inhibitors
* No concurrent warfarin
* No concurrent thiazide or loop diuretics
* No concurrent COX-2 inhibitors
* No concurrent NSAIDs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2003-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change in aromatase activity levels | From baseline to post-surgery

SECONDARY OUTCOMES:
Change in cell proliferation via a marker Ki67 between treatment arms by immunohistochemistry | From baseline to post-treatment
Correlation between aromatase activity and levels of COX 2 protein, HER 2/neu and ER status in surgical specimens | At post-treatment/surgery
Effect of treatment vs. no treatment on gene expression (mRNA) profile by microarray, kinase activities (PI3, AKT and ERK1/2 MAP kinases) and PGE2 levels | At post-treatment/surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Port, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States